CLINICAL TRIAL: NCT00696904
Title: Study of ABT-333 in Both Healthy Volunteers and Hepatitis C Virus (HCV) + Genotype 1 Infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Daniel Cohen, MD, Study Medical Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: M10-351
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2010-09

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — dasabuvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Other): Healthy volunteers, receiving 10-1200 mg ABT-333 or placebo, single dose
  Interventions: Drug: ABT-333; Drug: Placebo
- 2 (Other): HCV+ treatment-naive subjects receiving 100-300 mg ABT-333 or placebo, multi-dose, QD or BID
  Interventions: Drug: ABT-333; Drug: Placebo
- 3 (Other): Healthy volunteers, receiving 100 mg ABT-333, multi-dose, food effect
  Interventions: Drug: ABT-333

INTERVENTIONS:
Drug: ABT-333 — Capsule, see arms for intervention description
Drug: Placebo — Capsule, see arms for intervention description
  Arms: 1; 2

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics of ABT-333 in healthy volunteers and the antiviral activity in HCV infected subjects.

DETAILED DESCRIPTION:
Phase 1, double-blind, randomized, placebo-controlled clinical trial in healthy and HCV genotype 1 infected adults to evaluate safety, tolerability, antiviral activity and pharmacokinetics of ABT-333.

ELIGIBILITY:
Inclusion Criteria:

* Main Selection Criteria for Healthy Volunteers:

  * Subject has provided written consent.
  * Subject is in general good health.
  * If female, subject is postmenopausal.
  * If female, subject is not pregnant and is not breast-feeding.
* Main Selection Criteria for HCV+ Subjects:

  * Subject is HAV-IgM, HBsAg or HIV Ab negative.
  * Subject is HCV genotype 1 with HCV RNA of > 50,000 IU/mL.
  * Subject is excluded if they have previously received antiviral therapy for HCV infection
  * Subjects must demonstrate chronic hepatitis C infection for at least 6 months prior to study enrollment
  * Subjects must have a prior liver biopsy with histology consistent with HCV induced liver damage, and with no evidence of cirrhosis or liver pathology due to any cause other than chronic HCV.

Exclusion Criteria:

See above for main selection criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Analysis of pharmacokinetic variables and mean change in HCV RNA level from baseline. | approximately 1 week or less
Analysis of safety measures, including but not limited to tabulation of adverse events, physical exam, clinical lab results (include chemistry, hematology and urine) and vital signs. | approximately 1 week

SECONDARY OUTCOMES:
Analysis of variance of pharmacokinetic variables for subjects fasting or nonfasting. | approximately 1 week

REFERENCES:
- [Result] Mensing S, Polepally AR, Konig D, Khatri A, Liu W, Podsadecki TJ, Awni WM, Menon RM, Dutta S. Population Pharmacokinetics of Paritaprevir, Ombitasvir, Dasabuvir, Ritonavir, and Ribavirin in Patients with Hepatitis C Virus Genotype 1 Infection: Combined Analysis from 9 Phase 1b/2 Studies. AAPS J. 2016 Jan;18(1):270-80. doi: 10.1208/s12248-015-9846-1. Epub 2015 Nov 23. PMID 26597291